CLINICAL TRIAL: NCT03156881
Title: Global Osteopathic Treatment for Patients With Non-Alcoholic Fatty Liver Disease
Brief Title: Global Osteopathic Treatment for Patients With NAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jenna Wilcox (Other)
Responsible Party: Sponsor-Investigator, Jenna Wilcox, Thesis writer (Completed the 5 year osteopathic program), Canadian College of Osteopathy
Organization: Canadian College of Osteopathy (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCOsteopathy
Record Dates: First submitted 2017-05-12; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: 24 participants in control group receiving no global osteopathic treatment. Just standard care, baseline blood work every three months, improving their diet and exercise. They will also complete two questionnaires to measure their quality of life and readiness to change.
  Experimental group will also do the above with additional four osteopathic treatments to compare the differences in quality of life and liver function in both groups.
Who Masked: Participant
Masking Description: Since this study does not involve a sham treatment, the researcher and Dr. Peltekian have decided to have two consent forms. Patients will be assigned a code number and will be divided randomly into treatment or non-treatment groups via Dr. Peltekian opening up sealed envelops made by researcher Jenna Wilcox. Part one of the study will involve Dr. Peltekian asking potential participants consent to be a part of a study measuring " Quality of life and readiness for management of NAFLD". Upon consent, he/she will fill out the two questionnaires and give consent that their routine blood work can be analysed anonymously. During the same time, Dr. Peltekian will open up a sealed envelope revealing a code number and either an invitation to Part 2 of the study or not to invite and to remain as a control participant. By using this method the control group is not informed of the osteopathic research of the study (Part 2), thus reducing bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The participants in the treatment group (anticipating 24) will be receiving four global osteopathic treatments in a six week period alongside their standard care. Their standard care is to improve diet and increase exercise.Blood work done about every 3 months to check liver enzyme levels to observe improvements or monitor severity of the disease.
  This group will also complete questionnaires evaluating their quality of life (CLDQ) and their readiness to change before and after the treatment series.
  Interventions: Other: Global Osteopathic Treatment
- Control Group (No Intervention): This group will have an anticipated 24 participants and will continue their standard care as explained above along with completing two questionnaires evaluating their quality of life and readiness to change. This group will not be receiving any osteopathic treatment.

INTERVENTIONS:
Other: Global Osteopathic Treatment — The study objectives is to observe a difference and improvement of liver function based on liver enzyme count from blood work after osteopathic treatments. Also to observe an improvement in the patients quality of life after receiving treatment and in their readiness to change.
  Osteopathy is a type of manual therapy that uses gentle manipulations taking into consideration of the whole person when treating. For example if the liver is being treated, osteopaths look for mobility, to carry out its proper function. However one will also assess its interrelationships that can influence the liver such as its neighbours, articulating structures, example the diaphragm as well as its neurological input from T5-T9 for instance.
  Arms: Treatment group

SUMMARY:
Non-alcoholic fatty liver disease is a complex disease that is growing more prominent around the world especially in North America because of high prevalence of overweightness and obesity. There are many factors that are associated with this illness and it does not seem to be the same in every patient. The progression of this disease can with time lead to liver cirrhosis and even primary liver cancer (hepatocellular carcinoma). Currently, the only treatment plan involves diet change and exercise.

The goal of this research is to validate that Osteopathy can optimise patient health and to potentially be another option in preventing/reducing progression of this disease. This research is important for the future of Osteopathy to educate the public and other therapists/physicians the benefits this manual therapy has to offer. Previous research has been done and shown that Osteopathy can help patients with low back pain and type two diabetes, by affecting glucose and insulin levels with manipulation of the spine and pancreas.

Another study compared one group of obese patients with chronic low back pain that just did specific exercises to another group that were given exercises as well as Osteopathic manual therapy (OMT). Results showed both groups had reduced pain, however only the group with additional OMT showed improved range of motion in the thoracic spine, and showed greater degree of improvement overall for these patients. This study shows how OMT can be effective for individuals with NAFLD for in general these patients are obese and part of their treatment regime is to exercise to lose weight. The researcher could not find any previous research on OMT contributing to weight loss, however according to the Reve Pavilion natural health clinic website (2015), OMT can improve underlying issues such as low back pain, preventing the person to exercise effectively. The researcher also hopes to gain further knowledge of this subject, and to show the benefits of collaborating Osteopathy and Allopathic medicine together to obtain optimal patient care.

DETAILED DESCRIPTION:
Randomized Quantitative Clinical Trial. There will be 48 participants randomly assigned codes numbers and placed into a treatment group or non treatment group with 24 candidates in each. The control group will not be receiving treatments whereas the experimental group will be receiving four global osteopathic treatment over a six week period. All participants in both groups will have a baseline blood work provided by Dr. Peltekian a month before commencement of treatment. These patients have routine blood work every three months to begin with so they will get their second bloodwork done after the treatment sessions.

Each group will also fill out the Chronic liver disease questionnaire to measure quality of life and the URICA to measure their readiness to change a week before the first treatment, and a week after the last treatment session.

The study objectives is to observe a difference between blood work pre and post treatment that osteopathy has influenced and improved liver function based on liver enzyme count. Also to observe an improvement in the patients quality of life after receiving treatment and in their readiness to change. The researcher hopes to validate osteopathy as another treatment option to give NAFLD patients.

ELIGIBILITY:
Inclusion Criteria:

* Has a confirmed NAFLD diagnosis from Dr. Peltekian.
* Patient is abstaining from alcohol or consuming less than 20 g/day.
* Patient is willing to improve their lifestyle, diet and increase exercise.
* Patient can comprehend English for signing of consent forms.
* Agrees to abstain from any other type of manual therapy besides the researcher's osteopathic treatment during the study period.

Exclusion Criteria:

* Any other forms of liver disease. --> The current researcher is interested in a specific liver disease, NAFLD.
* Any tumors/cancer.--> The researcher does not want to interfere with cancer treatments. As well as the focus of this study is specifically how osteopathy can help patients with NAFLD, not patients with NAFLD plus cancer (more variables to deal with here).
* Patients with any psychiatric issues or dementia.--> Need proper consent to be able to do the study. Also participants need to be able to remember and compare the difference in how they truly feel before and after treatments on their quality of life that is being measured.
* Aneurysms/thrombosis. --> The researcher will be doing manual therapy on the body and is planning on working on the fluid/lymph level at times to decrease inflammation. The researcher wants the patient to be safe.
* Any patient abusing alcohol or any illicit drugs. --> The study is on NON-alcoholic fatty liver disease...not alcoholic.
* Any cardiovascular disease and Type 1 diabetes. --> Again researcher is trying to focus on the one liver disease NAFLD.
* Extremely high levels of Y glutamyltransferase (GGT): Normal range is: 8 to 65 U/L for adults. --> This will help to differentiate between NAFLD and alcoholic fatty liver disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-11 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Global osteopathic treatment will improve liver function in patient's with non-alcoholic fatty liver disease. | 6 weeks to complete treatment series. Approximately 12 weeks to receive all relative information to assess.
  Baseline blood work will be taken by Dr.Peltekian prior to commencement of treatments a month beforehand. Four osteopathic treatments will be given within a 6 week period. Then another blood sample will be given by Dr. Peltekian used to compare the differences from the baseline. The researcher will observe any change in liver enzymes, blood count, triacylgylceride levels from the previous blood work and with the control groups. The goal is to see an improvement of liver function from osteopathic treatments.
Global osteopathic treatment will increase quality of life in patients with non-alcoholic fatty liver disease. | Approximately 12 weeks.
  A Chronic Liver Disease Questionnaire( CLDQ) will be given to both control and treatment groups at the very beginning of the study ( first visit with Dr. Peltekian) and after the treatment series when getting their second blood work. The chronic liver disease questionnaire will be used and measured by Beth Bruce (statistician in Halifax Nova Scotia) using the Analysis of Variance. Data will be analyzed to detect differences over time, between groups and to determine if groups behave differently over time with respect to measures of quality of life. (ANOVA).
Global osteopathic treatment will increase readiness to change in patients with Non-Alcohoic Fatty Liver Disease using the URICA questionnaire. | Approximately 12 weeks.
  The University Rhode Island Change Assessment Scale(URICA) will be used to measure each patient's readiness to change ( to improve diet and exercise) in both groups. It will be given twice, a month before and after treatment series to see if osteopathic treatments will have an impact on a person's readiness to change.

CONTACTS AND LOCATIONS:
Overall Officials: Kevork Peltekian, MD, FRCPC, Principal Investigator — Division of Digestive Care & Endoscopy , Department of Medicine , Department of Surgery

IPD SHARING:
Plan to Share IPD: Undecided
Data sets that will be shared is anonymous blood work comparisons before and after osteopathic treatments to compare differences in a persons physiology. Also the results of the questionnaires given. Data will be only obtained if given permission from Dr.Kevork Peltekian and Jenna Wilcox.